CLINICAL TRIAL: NCT04269759
Title: Oral State and Knowledge, Attitudes and Practices of Pregnant Women on Their Oral Health and That of Their Unborn Child
Brief Title: 145/5000 Oral State and Knowledge, Attitudes and Practices of Pregnant Women on Their Oral Health and That of Their Unborn Child
Acronym: BUCCOMATER
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/14
Record Dates: First submitted 2020-02-07; First posted 2020-02-17 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Dental Care
Keywords: prevention; dental care; pregnancy
MeSH Terms: interventions — Surveys and Questionnaires; Dental Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnancy women
  Interventions: Other: Survey; Other: dental care

INTERVENTIONS:
Other: Survey — pregnant women will answer to a survey regarding their oral health knowledge, attitudes and practices for themselves and their unborn child
Other: dental care — pregnant women will have a dental care

SUMMARY:
Pregnancy is a physiological condition which is accompanied by changes in the oral sphere which may increase the need for oral care and prevention. The role of dental surgeons is to provide appropriate care and to provide information on the prevention of oral diseases of pregnant women but also of their unborn baby.

Investigators wants to determine if pregnants women know that national health insurance has set up a free dental care preventive examination.

DETAILED DESCRIPTION:
Investigators will describe the knowledge, attitudes and practices of pregnant women consulting at the maternity of Bordeaux University Hospital with regard to the oral examination of health insurance.

This study will also Evaluate the care needs and the acceptability of oral screening and study the association between the use of prenatal health insurance and dental health.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women

Exclusion Criteria:

* Patient refuses to participate in the study.
* Persons under guardianship
* No understanding of oral French.
* People with decompensated severe psychiatric disorder or severe cognitive impairment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Use of prenatal health insurance for free dental examination | Enrollment
  The use of this dental examination will be assessed with a survey

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France